CLINICAL TRIAL: NCT02418507
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Study to Evaluate the Effectiveness of a Proprietary Probiotic Blend on Functional Constipation
Brief Title: An Evaluation of the Effectiveness of a Proprietary Probiotic Blend on Functional Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: UAS Labs LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 14PPHU
Record Dates: First submitted 2015-03-06; First posted 2015-04-16 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Functional Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proprietary Probiotic Blend (Active Comparator): A proprietary probiotic blend: Lactobacillus acidophilus, Bifidobacterium lactis, Bifidobacterium longum, and Bifidobacterium bifidum at 56.75 mg
  Interventions: Dietary Supplement: Proprietary Probiotic Blend
- Placebo (Placebo Comparator): The placebo is administered to randomized healthy participants
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Proprietary Probiotic Blend — A proprietary probiotic blend: Lactobacillus acidophilus, Bifidobacterium lactis, Bifidobacterium longum, and Bifidobacterium bifidum at 56.75 mg
  Arms: Proprietary Probiotic Blend
Other: Placebo — The placebo is administered to randomized healthy participants
  Arms: Placebo

SUMMARY:
The primary objective for this study is to monitor the change in patient assessed symptoms of constipation in subjects taking the proprietary probiotic blend compared to those taking the placebo. The secondary objective for this study is to additionally monitor changes in stool consistency, stool frequency, quality of life and microbial composition of feces from baseline to Day 29, in all subjects. Safety considerations monitored any changes in blood safety parameters as well as incidence of adverse events throughout the entire study for all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults, aged 18 to 65 years
* BMI of 18.5 kg/m2 to 35.0 kg/m2 (inclusive)
* Subject is not of child bearing potential. Defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation) OR Female subject of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include:
* Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
* Double-barrier method (condoms with spermicide or diaphragm with spermicide)
* Non-hormonal intrauterine devices
* Vasectomy of partner
* Non-heterosexual lifestyle
* Subjects must have at least two of the following criteria based on subject self-reporting, for the past 3 months with the symptoms beginning at least 6 months ago:
* Two or more criteria must be met by subjects:

  1. Straining during at least 25% of defecations
  2. Lumpy or hard stools in at least 25% of defecations
  3. Sensation of incomplete evacuation for at least 25% of defecations
  4. Sensation of anorectal obstruction/blockage for at least 25% of defecations
* Fewer than three defecations per week
* Loose stools are rarely present without the use of laxatives
* Insufficient criteria for Irritable Bowel Syndrome
* Subjects with an average stool type of < 3 on the Bristol Stool Scale as assessed over the two week run-in period (confirmed at baseline review of bowel habits diary).
* Subjects who agree to maintain their current level of physical activity throughout the trial period.
* Subjects who agree to discontinue the use of probiotic supplements including foods supplemented with probiotics (i.e. yogurts) or fiber supplements including foods labeled as supplemented with fiber
* Subjects who agree to discontinue use of over-the-counter laxative medications (other than the rescue medication provided) within 2 weeks of screening and throughout the trial.
* Subjects who successfully complete the run-in period by completing at least 80% of Run-In diary entries, 100% of IPAQ questionnaires and provide fecal sample.
* Subjects who understand the nature and purpose of the study including the potential risks and side effects
* Subjects who are willing to complete all study procedures including study related questionnaires and comply with study requirements
* Subjects who have given voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

* Subjects who are pregnant, breastfeeding or planning on becoming pregnant throughout the course of the study.
* Subjects with any unstable medical conditions
* Subjects with any major diseases of the cardiovascular, renal, hepatic, gastrointestinal, pulmonary or endocrine systems
* Subjects with Type I or Type II diabetes
* Subjects with a history of major gastrointestinal complications (i.e. Crohn's disease, ulcer, cancer, ulcerative colitis)
* History of or current diagnosis of any cancer (except for successfully treated basal cell carcinoma) diagnosed less than 5 years prior to screening. Subjects with cancer in full remission more than 5 years after diagnosis are acceptable
* Subjects with neurological disorders or significant psychiatric illnesses (significance determined by the Qualified Investigator)
* Subjects who are immuno-compromised (HIV positive, on anti-rejection medication, rheumatoid arthritis)
* Subjects with any medical condition or a history of abdominal surgery that is deemed exclusionary by the Qualified Investigator
* Subjects who have features which may suggest a more serious underlying cause of chronic constipation such as rectal bleeding, anemia, abrupt weight loss ( 5kg or more within the past month prior to randomization), gastrointestinal polyps, first degree family history of colorectal cancer.
* Subjects with an active eating disorder
* Subjects who have used an over-the-counter or prescription laxative medication within 2 weeks prior to screening.
* Subjects who have used probiotic or fiber supplements (or probiotic/fiber enriched foods) within 4 weeks prior to screening
* Subjects who have used an antibiotic within 4 weeks prior to screening
* Subjects who have used medications in the investigators opinion known to cause constipation (i.e. opiates) within 4 weeks of screening
* Subjects using Medicinal Marijuana
* Subjects who use illicit drugs or have a history of alcohol or drug abuse within the past 6 months
* Subjects who currently consume greater than 2 standard alcoholic drinks per day.
* Subjects who have participated in a clinical research trial within 30 days prior to randomization.
* Subjects with an allergy or sensitivity to the investigational product ingredient
* Subjects who are cognitively impaired and/or who are unable to give informed consent
* Subjects who have abnormal laboratory results or any other medical or psychological condition which, in the opinion of the Principle Investigator, may adversely affect the subjects' ability to complete the study or its measures or which may pose significant risk to the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-05-29 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Changes in the symptoms of constipation as measured by the PAC SYM questionnaire | Baseline to Day 29

SECONDARY OUTCOMES:
Changes in stool consistency as measured by the Bristol Stool Scale | Baseline to Day 29
Changes in stool frequency | Baseline to Day 29
  Weekly mean Complete Spontaneous Bowel Movements
Changes in quality of life questionnaire score | Baseline to Day 29
Changes in microbial composition of feces | Baseline to Day 29

OTHER OUTCOMES:
Changes in blood safety parameters | Baseline to Day 29
  CBC, electrolytes, creatinine, AST, ALT, GGT and bilirubin

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Pelipyagina, MD, Principal Investigator — tetyana@kgksynergize.com
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada